CLINICAL TRIAL: NCT01879111
Title: Increasing the Efficiency of Depression-screening Using Patient-targeted Feedback: Randomized Controlled Trial
Brief Title: Increasing the Efficiency of Depression-screening Using Patient-targeted Feedback
Acronym: DEPSCREEN-INFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: 01-GX-1004; DRKS00003277 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2013-06-12; First posted 2013-06-17 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Depressive Episode; Chronic Ischaemic Heart Disease; Hypertension
Keywords: Depressive episode; Chronic ischaemic heart disease; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- state-of-art depression screening + patient-targeted feedback (Experimental): Using a randomised-controlled study design half of the patients will receive a patient-targeted written screening feedback. This feedback contains information about depression in general, depression-severity adapted treatment guidelines and contact-information for treatment.
  Interventions: Other: patient-targeted feedback
- state-of-art depression screening (No Intervention)

INTERVENTIONS:
Other: patient-targeted feedback — Using a randomised-controlled study design half of the patients will receive a patient-targeted written screening feedback. This feedback contains information about depression in general, depression-severity adapted treatment guidelines and contact-information for treatment.
  Arms: state-of-art depression screening + patient-targeted feedback

SUMMARY:
Out-patients with coronary heart disease or hypertension will fill out a depression screening questionnaire while waiting in a cardiac clinic. Using a randomised-controlled study design half of the patients will receive a patient-targeted written screening feedback. This feedback contains information about depression in general, depression-severity adapted treatment guidelines and contact-information for treatment. Patients in the control group receive no direct screening-feedback but their cardiologist will be informed about the screening result. All patients with a positive screening-result will be contacted after one month and six months and asked for symptoms of depression, and their use of health care. The aim of this study is to evaluate the efficiency of this minimal intervention on the course of depressive symptom in patients with known coronary heart disease or hypertension.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficiency of a minimal intervention on the course of depressive symptoms in patients with known coronary heart disease (CHD) or hypertension. By means of a depression screening and individual patient-targeted feedback the level of depression should decrease, the percentage of treated depressed patients should increase and health economic costs should be lowered. The main hypothesis is that screening plus targeted feedback results in a greater reduction of depression than screening only.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Both, male and female
* Minimum Age: 18 Years
* Maximum Age: no maximum age
* Attendance in a cardiac clinic;
* Clinical diagnosis of coronary heart disease or hypertension;
* Age ≥ 18 years;
* Sufficient language skills;
* Informed consent

Exclusion Criteria:

* Life threatening health status;
* Severe somatic or/and psychological disorder that needs urgent treatment;
* Acute suicidal tendency;
* Severe cognitive or/and visual difficulties;
* Not being able to fill out questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4151 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Level of depression one month after screening (Patient Health Questionnaire-9) | One month after depression screening

SECONDARY OUTCOMES:
Level of depression six months after screening (Patient Health Questionnaire-9) | One month and six months after screening
Proportion of patients treated for depression. | One month and six months after screening
Direct and indirect health costs | One month and six months after screening
Quality-adjusted years of life and quality of life (EuroQol-5D) | One month and six months after screening

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Loewe, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (2):
- Germany (2):
  - University Medical Center Universitaeres Herzzentrum Hamburg-Eppendorf, Hamburg
  - Cardiologicum Hamburg, Hamburg

REFERENCES:
- [Derived] Lowe B, Blankenberg S, Wegscheider K, Konig HH, Walter D, Murray AM, Gierk B, Kohlmann S. Depression screening with patient-targeted feedback in cardiology: DEPSCREEN-INFO randomised clinical trial. Br J Psychiatry. 2017 Feb;210(2):132-139. doi: 10.1192/bjp.bp.116.184168. Epub 2016 Dec 1. PMID 27908896
- See also: Website of the Department of Psychosomatic Medicine (in German) — https://www.uke.de/kliniken-institute/kliniken/psychosomatische-medizin-und-psychotherapie/forschung/arbeitsgruppen/ag_koerperliche-erkrankungen.html